CLINICAL TRIAL: NCT04400786
Title: A Randomized Open-labeled Study for Comparison of Patient-reported Outcomes Between Two Therapeutic Schedules of Imrecoxib in Ankylosing Spondylitis
Brief Title: A Randomized Open-labeled Study for Comparing Methods of Using Imrecoxib to Treat AS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Wu Jieping Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AROS-MIAS
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Ankylosing Spondylitis; Therapeutic Agent Toxicity
MeSH Terms: conditions — Spondylitis, Ankylosing; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Intervention Model Description: Patients were randomly divided into the continuous treatment group and the on-demand treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- On-demand treatment (Experimental): This group of 98 ankylosing spondylitis patients is prescribed with intermittent Imrecoxib (100mg.prn.po) according to the feeling of pain till 24 weeks. The sulfasalazine (500mg.tid.po) is used.
  Interventions: Procedure: intermittent treatment
- Continuous treatment (Active Comparator): This group of 98 ankylosing spondylitis patients is prescribed with continuous Imrecoxib (100mg.bid.po) for 24 weeks. The sulfasalazine (500mg.tid.po) is used.
  Interventions: Procedure: continuous treatment

INTERVENTIONS:
Procedure: intermittent treatment — According to the feeling of pain, the on-demand treatment group is prescribed with or without Imrecoxib (100mg/tablet, 100mg.prn.po), but the maximal dose does not exceed 100 mg per time, twice (morning and evening) per day. The duration lasted for 24 weeks.
  Arms: On-demand treatment
Procedure: continuous treatment — The continuous treatment group is prescribed Imrecoxib (100mg.bid.po) regardless of the pain in the treatment course for 24 weeks.
  Arms: Continuous treatment

SUMMARY:
The selective cox-2 inhibitor has been widely used in the treatment of Ankylosing spondylitis (AS). The Imrecoxib is a new cox-2 inhibitor. But the treatment strategy has not been decided yet. To determine which is better in treating AS in the methods between on-demand treatment and continuous treatment. To solve this question, we designed this study.

DETAILED DESCRIPTION:
Ankylosing spondylitis (AS) is a chronic systemic inflammatory arthritis of unknown etiology, occurring in young men aged 16-25 and presenting the genetic predisposition. AS is a common rheumatic disease, with a prevalence of 0.3 ~ 0.5% in general people of China, which means that about 5 million people in our country suffer from this disease. AS mainly invades the central axis, characterized by the inflammation of sacroiliitis and attachment points. The onset of AS is insidious. The early clinical manifestations are mainly inflammatory low back pain, which gradually affects the lumbar spine, thoracic vertebrae, and cervical vertebrae. The persistent inflammation will gradually stiffen and fuse the joints, causing osteoporosis and destruction of the vertebral body, resulting in the ossification of ligaments, and leading to the disability ultimately. Except for the joint lesions, AS is usually accompanied by multiple extra-articular manifestations, such as uveal inflammation, psoriasis, inflammatory bowel disease, etc. Especially, AS is often complicated with multiple complications symptoms, such as arthritis, arterial disease, fibromyalgia, depression, etc. In summary, AS has seriously affected the normal work and work of patients, which has become the main reason for the labor loss in young and middle-aged people. Therefore, it is of great value for controlling inflammation effectively and alleviate joint pain to improve the life quality of patients and save social labor.

Non-steroid anti-inflammatory drugs (NSAIDs), the anti-inflammatory and analgesic drugs and widely used in rheumatic diseases, can effectively relieve pain and quickly improve the symptoms of inflammatory joint disease. The role of NSAIDs in the treatment of AS is very important, which could not only generate anti-inflammatory effect, but also improve the joint function, delay joint erosion, and prevent the formation of osteophyte. The treatment guidelines of AS in American Rheumatology Association / American Spondyloarthropathy Collaboration in 2015 recommended continuous prescription NSAIDs as the first-line treatment for patients with active AS. In the 2016 ASAS / European Guideline of Axial Spondyloarthropathy, NSAIDs should be treated as the first-line treatment for patients with joint pain and joint stiffness. Those who respond well to NSAIDs are recommended for continuous treatment. The latest 2018 APLAR guidelines also recommend that NSAIDs should be used as first-line treatment for active AS, but the method of continuous treatment or treatment on demand is not discussed because two clinical trials have shown that the efficacy of on-demand is not worse than continuous treatment. In summary, NSAIDs are recommended for the first-line treatment of AS, but the differences in the efficacy, safety, and patient benefit between continuous treatment and on-demand treatment, as well as the treatment course, is controversial yet.

NSAIDs could inhibit the activity of cyclooxygenase (COX), blocking the conversion of arachidonic acid to prostaglandins, prostacyclin, and thromboxane A2. In addition, NSAIDs could also inhibit the release of bradykinin, inhibit lymphocyte proliferation, and reduce the migration of granulocyte and macrophages in inflammation. COX includes COX-1 and COX-2. COX-1 induced prostaglandins mainly generate the physiological and protective effect, such as maintaining the integrity of the gastrointestinal mucosa, adjusting the renal blood flow, and guarantee the function of platelets. COX-2 is mainly expressed in macrophages, fibroblasts, cartilage and endothelial cells with a low level in the basic state. Once stimulated by cytokines or endothelin, the expression will tremendously increase several times, induce the production of prostaglandins, and participate in inflammation. NSAIDs could be classified as non-specific COX inhibitors, selective COX-1 inhibitors, and selective COX-2 inhibitors based on the effects of different COX. The main adverse reaction of NSAIDs derives from its inhibitory effect on COX-1, causing adverse gastrointestinal reactions. And the gastrointestinal ulcers and bleeding are also the most common causes of hospitalization and death. The selective COX-2 inhibitor is the new generation of NSAIDs, with better anti-inflammatory and analgesic effects, in that it could specifically inhibit the COX-2 but has no effect on COX-1, greatly reducing the adverse reaction of gastrointestinal tracts and kidneys. Multiple clinical trials and meta-analysis have shown that selective COX-2 inhibitors can significantly reduce the gastrointestinal symptoms and peptic ulcer formation in the endoscopic. Therefore, selective COX-2 owns a much more general application space in rheumatic diseases.

Most of the COX-2 inhibitors in China are not original research drugs previously, and only Celecoxib is available in the United States according to FDA. Unearthing new selective cox-2 inhibitor is necessary. Imrecoxib is a COX-2 inhibitor designed by the Chinese Academy of Medical Sciences and Jiangsu Hengrui Hospital Co., Ltd. in China, which has been approved by the Chinese Food and Drug Administration (CFDA) for marketing. The recommended dose of Imrecoxib is 100mg. bid.po. according to the instructions. Studies in vitro has demonstrated that Imrecoxib could specifically inhibit the COX-2, and inhibit the expression of COX-2 mRNA to restrain the inflammation. Multiple clinical studies have demonstrated that Imrecoxib was effective in treating osteoarthritis, with similar efficiency to Celecoxib but without severe gastrointestinal adverse effect, with a lower percentage of cardiovascular adverse effect, and with relatively good safety. In 2017, the comparison between Imrecoxib and Celecoxib in treating serum-negative spondyloarthropathy (SPA) revealed that the effect of Imrecoxib (10mg.bid.po for 12 weeks) was not worse than that of Celecoxib, which could significantly alleviate disease activity, joint function and inflammatory markers. But there is a lack of study with a large sample size and long course to further demonstrate the effectiveness and safety of Imrecoxib in treating SPA and AS.

The AS disease activity score such as BASDAI and radiological assessment are the main observation indicators for efficacy evaluation in the clinical study of NSAIDs treating AS for the moment. But the evaluation of life quality is also important for patients with AS, which includes 4 respects, the body 's function, disease activity, economic status, and social status. Data from Taiwan shows that a variety of factors can affect the patient 's life quality except for the disease activity, including the course of the disease, drinking, weight, mental, and economic factors, etc. So, adequate life quality assessment and support should be given to the AS patients. However, there is a lack of studies that employed patients self-report and patients' life quality assessment as the main observation indicators. The present study intends to use the results of patients' self-report as the evaluation criteria, to compare the efficacy and safety between continuous treatment and on-demand treatment of Imrecoxib for AS under different treatment modes, which could also provide direct evidence for the optimized applications in rheumatic diseases.

Meanwhile, we also want to find whether on-demand treatment of Imrecoxib could reduce the occurrence of adverse reactions, reduce the economic burden, and bring more benefits under the premise that the on-demand treatment is not worse than continuous use of Imrecoxib in drug efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 ~ 65 (both ends included), regardless of gender;
2. The condition is in the active period, evaluation criteria: Bath Ankylosing Spondylitis-Disease Activity Index (BASDAI) ≥4 (scale 0-10cm);
3. ESR ≥20mm / h or hsCRP ≥3mg / L;
4. Naive patients who have not received any drugs or physical treatment to treat the AS; or patients who discontinued all therapeutic drugs for more than 3 months.
5. Female subjects with fertility must agree to take effective contraceptive measures in the trial.

Exclusion Criteria:

1. complicated with other rheumatic diseases, such as inflammatory bowel disease, psoriasis, active uveitis, rheumatoid arthritis, systemic lupus erythematosus, primary Sjogren's syndrome, systemic vasculitis, etc.
2. the anti-infection treatment due to the active periods of acute and chronic infections such as mycobacterium tuberculosis, hepatitis B, hepatitis C, HIV, etc.
3. complicated with the malignant tumor.
4. complicated with the drug allergies (including sulfonamides, NSAIDs, etc.), allergic diseases or allergies.
5. Pregnant or lactating women.
6. Abnormal blood system: hemoglobin <80g / L, white blood cells <4.0 × 109 / L, platelet < 100 × 109 / L.
7. Insufficient liver and kidney function: 1.5 times higher than the upper limit of normal value of ALT and AST; 1.25 times higher than the upper limit of normal value of creatinine and urea nitrogen.
8. Insufficient heart function: New York's heart association (NYHA) level ≥ grade II.
9. The usage of analgesic drugs (such as methadone, morphine, etc.) within 4 weeks before baseline.
10. Patients received the spine or joint surgery within 2 months before of the enrollment.
11. Patients participated the any other clinical trials within 3 months before of the enrollment.
12. Patients received live vaccination within 3 months before the enrollment.
13. Patients refused to sign the informed consent form, or the patient lack the capacity to decide for themselves.

Elimination criteria:

1. Violation of the diagnostic criteria for AS.
2. Serious violation of the trial, and the investigators believe that it is not feasible to exclude subjects who cannot be evaluated for effectiveness.
3. No follow-up records after the enrollment.

Exit criteria

1. The subjects request to stop using the experiment drug in the study.
2. Investigators believe that subjects should be withdrawn due to clinical adverse events.
3. The subject is pregnant.
4. Serious violation of the study protocol, which affects the effectiveness and safety evaluation.
5. The subject cannot or does not comply with the requirements of the research project.
6. Subjects who receive any surgical treatment in the study.
7. The investigators believe that further participation in the study is not consistent with the best interests of the subjects.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2020-05-07 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
The percent of subjects who achieved moderate improvement in SRM at the 24th week; | 24 weeks
  The indicator to evaluate the improvement of ASAS HI is the standardized response mean (SRM, SRM = mean / standard deviation the interval of ASAS HI before and after treatment), SRM <0.4 indicates mild improvement, SRM 0.4-0.79 indicates moderate improvement, SRM≥0.8 indicates severe improvement.The percent of patients who achieved moderate improvement in SRM at the 24th week is observed.

SECONDARY OUTCOMES:
The percent of subjects who achieved moderate improvement in SRM at the 12th week. | 12 weeks.
  The indicator to evaluate the improvement of ASAS HI is the standardized response mean (SRM, SRM = mean / standard deviation the interval of ASAS HI before and after treatment), SRM <0.4 indicates mild improvement, SRM 0.4-0.79 indicates moderate improvement, SRM≥0.8 indicates severe improvement. The percent of patients who achieved moderate improvement in SRM at the 12th week.
The percent of subjects who achieved severe improvement in SRM at the 12th week. | 12 weeks.
  The indicator to evaluate the improvement of ASAS HI is the standardized response mean (SRM, SRM = mean / standard deviation the interval of ASAS HI before and after treatment), SRM <0.4 indicates mild improvement, SRM 0.4-0.79 indicates moderate improvement, SRM≥0.8 indicates severe improvement. The percent of patients who achieved severe improvement in SRM at the 12th week is evaluated.
The percent of subjects who achieved severe improvement in SRM at the 24th week. | 24 weeks.
  The indicator to evaluate the improvement of ASAS HI is the standardized response mean (SRM, SRM = mean / standard deviation the interval of ASAS HI before and after treatment), SRM <0.4 indicates mild improvement, SRM 0.4-0.79 indicates moderate improvement, SRM≥0.8 indicates severe improvement. The percent of patients who achieved severe improvement in SRM at the 24th week is evaluated.
The change of self-evaluation compared with the baseline | 2, 4, 8, 12, 24 weeks.
  The slef-evaluation is performed with self-evaluation visual simulation method (0~40, higher score indicate more severe condition). The comparison was made between the baseline and the different time point in the follow-up.
The change of BASDI compared with the baseline. | 2, 4, 8, 12, 24 weeks.
  The disease activity was evaluated by the Bath Ankylosing Spondylitis Disease Activity Index (BASDI, 0~70, higher score indicates more severe condition). The comparison was made between the baseline and the different time point in the follow-up.
The relation between disease activity assessment and patient self-assessment | 12, 24 weeks.
  The correlation analysis between disease activity assessment (BASDI) and patient self-evaluation (self-evaluation visual simulation method).
Safety assessment including adverse effects such as gastrointestinal tract symptoms of two prescription strategy | 2, 4, 8, 12, 24 weeks.
  The safety assessment indicates the adverse effects or severe adverse effects in the follow-up including disability, prolonged hospitalization, death and so on.
The cost-effectiveness of two prescription strategy | 24weeks.
  The average cost-effectiveness ratio analysis of two prescription strategy was compared.

CONTACTS AND LOCATIONS:
Overall Officials: Lindi Jiang, PhD, Study Chair — Fudan University
Locations (1):
- Lindi Jiang, Shanghai, China

IPD SHARING:
Plan to Share IPD: No